CLINICAL TRIAL: NCT04050592
Title: Randomized Comparative Trial Between Abrupt and Tapered Discontinuation of Postmenopausal Hormone Therapy: Impact on Endothelial Function, Recurrence of Vasomotor Symptoms and Quality of Life
Brief Title: Discontinuation of Postmenopausal Hormone Therapy: Impact on the Cardiovascular System and Quality of Life
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanna Savolainen-Peltonen (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Sponsor-Investigator, Hanna Savolainen-Peltonen, M.D., Ph.D., associate professor, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: FINNHT1
Record Dates: First submitted 2019-06-18; First posted 2019-08-08 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Menopause; Atherosclerosis; Cardiovascular Diseases; Estrogen Replacement Therapy
Keywords: Randomized Controlled Trial; Menopause; Hormone Therapy; Vasomotor symptoms; Quality of Life; Cardiovascular diseases; Endothelium
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A, Abrupt Discontinuation (Other): Women in group A will discontinue HT (estradiol, 2 mg daily) abruptly after study week 9 and will continue with placebo for study weeks 10-20.
  Interventions: Drug: Estradiol; Other: Placebo
- Group B, Tapered Discontinuation (Other): Women in group B will discontinue HT (estradiol, 2 mg daily) gradually during study weeks 7-9, as follows:
  * weeks 7-9: 1 mg estradiol daily for 10 days and then 1 mg estradiol every other day for 11 days.
  * weeks 10-20: placebo
  Interventions: Drug: Estradiol; Other: Placebo
- Group C, Control Group (Active Comparator): Women in Group C, the control group, will continue with HT (estradiol, 2 mg daily) throughout the whole study period of 20 weeks.
  Interventions: Drug: Estradiol

INTERVENTIONS:
Drug: Estradiol — Active intervention is estradiol. Hormone therapy (HT) of all 150 participants will be standardized to 2.0 mg of oral estradiol (E2) without progestogen for six weeks prior to randomization. After that participants will be randomized into three groups (A, B, C) of equal size.
Other: Placebo — Those in groups A and B will switch from estradiol to placebo at the beginning of the 10th week after abrupt or tapered discontinuation of HT.
  Arms: Group A, Abrupt Discontinuation; Group B, Tapered Discontinuation

SUMMARY:
Although the impact of postmenopausal hormone therapy (HT) on cardiovascular disease risk has been studied in several large randomized trials, little is known about the acute cardiovascular consequences of HT discontinuation. In this randomized, double-blind, placebo-controlled trial, the investigators will compare the cardiovascular consequences of abrupt and tapered modes of HT discontinuation in 150 Finnish healthy postmenopausal women under age 60 years. The primary outcome is brachial artery flow-mediated dilatation. In addition, biochemical markers will be measured during the study period of 20 weeks. Health-related quality of life, frequency of hot flush recurrence and other menopausal symptoms will be also assessed in these groups. The trial will provide new high-quality information about the cardiovascular safety as well as the correct timing and method of HT discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* healthy postmenopausal women
* age ≤ 60 years
* has used postmenopausal hormone therapy for at least 3 years

Exclusion Criteria:

* any clinically significant disease
* use of regular medication
* history of cardiovascular events
* history of smoking
* body mass index over 30 kg/m2
* thickness of endometrium over 6 millimeters

Max Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation (FMD) | 8 and 14 weeks
  The primary outcome in this study is brachial artery flow-mediated dilation (FMD) to assess endothelial function. To induce reactive hyperemia, a sphygmomanometer cuff is placed on the forearm and inflated to a suprasystolic pressure for five minutes, after which the cuff is deflated. The brachial artery diameter is measured at baseline and during reactive hyperemia, and the relative change in diameter (in millimeters) is calculated. We measure FMD at baseline (at study week 5) and after HT discontinuation (at study weeks 13 and 19).

SECONDARY OUTCOMES:
Symptom diary | 5 and 13 weeks
  Participants will keep a symptom diary reporting the exact number, severity and timing of hot flashes during three periods each lasting three weeks: the first period at baseline, the second starting on the 10th week and the third starting on the 18th week. Based on the diary notes, we can assess, how frequent, severe and durable the symptoms are during each period.
Women's Health Questionnaire | 5 and 13 weeks
  Women's Health Questionnaire measures emotional and physical health. WHQ includes 37 questions that are answered based on the momentary feeling on a four-point scale (Yes, definitely; Yes, sometimes; No, not so much; No, not at all). The participant receives 37 points at minimum and 148 points at maximum.
Symptom questionnaire | 5 and 13 weeks
  The symptom questionnaire includes 19 questions about the frequency of menopausal symptoms (such as hot flashes, night sweats and insomnia) experienced during the past two weeks, and each question is evaluated on a four-point scale (never or seldom; once a month; once a week; almost daily).The participant receives 19 points at minimum and 76 points at maximum.
European Quality of Life Instrument | 5 and 13 weeks
  EuroQoL includes a health classification index that covers five dimensions of HRQL (mobility, self-care, usual activities, pain/discomfort, anxiety/depression).The participant receives 5 points at minimum and 15 points at maximum.
  In the second part of the questionnaire, there is a visual analogue scale ranging from 0, "worst imaginable health state", to 100, "best imaginable health state". Thus, the participant receives from 0 to 100 points from this part of the questionnaire.
Female Sexual Function Index | 5 and 13 weeks
  This questionnaire includes 19 questions about sexuality. The questions are answered on a five-point scale (almost always or always; most times; sometimes; a few times; almost never or never). The participant receives 19 points at minimum and 95 points at maximum.
Biomarker: Concentration of endothelin-1 | 5 and 8 weeks
  Concentration of endothelin-1 (ET-1, a vasoconstrictive marker, unit pmol/l)
Biomarker: Concentration of nitrite and nitrate | 5 and 8 weeks
  Concentration of nitrite and nitrate (markers of released nitric oxide and consequent vasodilation, unit µmol/l)
Biomarker: Concentration of Asymmetric Dimethylarginine | 5 and 8 weeks
  Concentration of asymmetric Dimethylarginine (ADMA, inhibitor of NO synthesis and indicator of endothelial dysfunction, unit µmol/l)
Biomarker: concentration of sex hormones | 2, 5 and 8 weeks
  Concentration of sex hormones: Follicle-stimulating hormone (FSH, unit IU/l), luteinizing hormone (LH, unit IU/l), estrone (pmol/l), estradiol (nmol/l) and sex hormone-binding globulin (SHBG, unit nmol/l)
Biomarker: Concentration of coagulation factors | 5 and 8 weeks
  Concentration of coagulation factors: fibrinogen (g/l), plasminogen activator inhibitor-1 (IU/ml), D-dimer (mg/l)
Biomarker: Concentration of lipids | 5 and 8 weeks
  Concentration of lipids: high-density lipoprotein cholesterol (HDL, unit mmol/l), low-density lipoprotein cholesterol (LDL, unit mmol/l), very low-density lipoprotein cholesterol (VLDL, unit mmol/l), triglycerides (mmol/l) and lipoprotein A (g/l)
Biomarker: Concentration of carbohydrate metabolism | 5 and 8 weeks
  Concentration of carbohydrate metabolism: fasting glucose (mmol/l) and insulin (mU/l)
Biomarker: Concentration of oxidative stress | 5 and 8 weeks
  Concentration of oxidative stress: oxidized LDL (U/l)
Biomarker: Concentration of inflammatory factors | 5 and 8 weeks
  Concentration of interferon-γ (IFN-γ, unit ng/ml), monocyte chemoattractant (MCP-1, unit pg/ml), macrophage inflammatory protein 1α (MIP-1α, unit pg/ml), tumor necrosis factor α (TNF-α, unit pg/ml) and high-sensitivity C-reactive protein (hs-CRP, unit mg/l)
Biomarker: Concentration of advanced glycation end products and soluble form of their receptor | 5 and 8 weeks
  Concentration of advanced glycation end products (AGE, unit U/ml) and soluble form of their receptor (sRAGE, unit pg/ml)
Biomarker: Concentration of cellular adhesion molecules | 5 and 8 weeks
  Concentration of cellular adhesion molecules: E selectin (mg/dl), intracellular cell-adhesion molecule-1 (ICAM-1, unit ng/ml), vascular cell adhesion molecule-1 (VCAM-1, unit ng/ml)
Concentration of matrix metalloproteinases | 5 and 8 weeks
  Concentration of matrix metalloproteinases (MMPs, unit µM)
Rey Auditory Verbal Learning Test (RAVLT) | 1 and 19 weeks
  RAVLT evaluates a wide diversity of cognitive functions. Participant is given a list of 15 unrelated words repeated over five different trials and are asked to repeat. Another list of 15 unrelated words are given and the client must again repeat the original list of 15 words and then again after 30 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Tomi Mikkola, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- HUS Women's Hospital, Helsinki, Finland